CLINICAL TRIAL: NCT06530056
Title: Effects of Costovertebral Mobilization on Kyphotic Posture and Lung Function in Non Smoker
Brief Title: Costovertebral Mobilization on Kyphotic Posture and Lung Function in Non-Smoker
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rida Mumtaz
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Hyperkypohsis and Impaired Lung Function
Keywords: Hyperkyphosis; Pulmonary Functions; Costoverterbral Mobilization; FEV1/FVC; Cobb Angle
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Costovertebral Mobilization+Conventional Therapy (Experimental): Costovertebral mobilization:
  It will be performed in 3 Different Positions to target specific regions of rib cage.
  Conventional Therapy:
  Hot pack 10 mints, Posture corrective exercises, Breathing exercises.
  Interventions: Other: Costovertebral Mobilization+Conventional Therapy
- Conventional Therapy (Other): Conventional Therapy:
  Hot pack 10 mints, Posture corrective exercises, Breathing exercises
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Costovertebral Mobilization+Conventional Therapy — Patient would receive costovertebral mobilization in side lying position for left 10th to 6th, in sitting position for right 10th to 2nd rib and in supine lying position for 1st rib.
  Conventional Therapy:
  Hot pack 10 mints, Posture corrective exercises, Breathing exercises Frequency; 4 times/week for 3 weeks
  Arms: Costovertebral Mobilization+Conventional Therapy
Other: Conventional Therapy — Electrotherapy:
  • Hot Pack 10 minutes
  Posture Corrective Exercises:
  * Thoracic Rotation 10 rep/session
  * Thoracic extension 10 rep/session
  * Scapular retraction 5 rep/session
  * Deep neck flexor Isometric 5 rep/session
  Deep Breathing Exercises:
  • Pursed lip breathing 10 repetition in one session
  Arms: Conventional Therapy

SUMMARY:
Aim of this study is to find the effects of Costoverterbral Mobilization on Thoracic kyphosis and Lung function in non-smoker. A randomized control trial that will include total 44 participants.The first group will receive Costovertebral Mobilization along with conventional therapy and 2nd group will receive conventional therapy.Data collected will be analyzed through SPSS 25

DETAILED DESCRIPTION:
Kyphosis is the curvature of the thoracic spine, formed by the shape of the vertebrae and the intervertebral discs and-in standing position-paraspinal muscle strength. Hyperkyphosis is usually associated with increased anteroposterior diameter of the thorax and a decrease in the distance between the xiphisternum and pubis and it is present when the kyphosis angle exceeds the normal ranges. This curve is concave anteriorly with a normal angle between 20˚ - 40˚.

The lungs are the foundational organs of the respiratory system,whose most basic function is to facilitate gas exchange from the environment into the bloodstream.The decline in lung function could be associated with hyperkyphosis, As the curvature of the thoracic spine increases and the posture becomes more hunched, the mobility of the rib cage could be limited and restrict the thoracic and lung expansions during inspiratory maneuver.

Different treatment strategies such as surgery, splinting, exercises and manual therapies such as massage, muscle energy technique, and passive joint mobilization have been used to treat hyperkyphosis. Costovertebral mobilization is a manual therapy technique, to improve the mobility and function of the joints between the ribs (costo) and the vertebrae (vertebral). This technique increases the range of motion of ribcage and spine, thus improve kyphosis posture and lung functions.

ELIGIBILITY:
Inclusion Criteria:

* Non smoker
* Age: 20-40 years
* Normal Body Mass Index 18.5 To 24.9
* Both female and male gender
* Decrease forced expiratory volume-one second/ forced vital capacity ratio greater than or equal to 70%
* Increase Thoracic kyphotic posture greater than or equal to 40˚

Exclusion Criteria:

* Any respiratory disease of the upper or lower respiratory tracts e.g. asthma, chronic bronchitis, COPD, emphysema etc. which could altered the optimal lung functioning.
* Previous history of rib fractures, dislocations, sprains of costochondral, costosternal and interchondral joints.
* Smokers
* Scheuermann Disease
* Primary and Secondary neoplastic lesions of the spine and/or ribs
* Obvious advanced spinal deformity e.g. kyphoscoliosis
* Infection e.g. tuberculosis
* Primary and secondary neoplastic lesions of the soft tissue structures of the chest
* Inflammation e.g. acute rheumatoid arthritis or ankylosing spondylitis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
X-RAY | 3 weeks
  X-ray is a gold standard method for objective assessment of Thoracic Kyphosis.

SECONDARY OUTCOMES:
Spirometer | 3 weeks
  For measurement of forced expiratory volume-one second/ Forced vital capacity ratio (Pulmonary Function Tests).

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Ali, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Madiha Ali, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No